CLINICAL TRIAL: NCT04069117
Title: Follicular Synchronization in Polycystic Ovarian Syndrome Patients Undergoing Intracytoplasmatic Sperm Injection With Letrozole /Antagonist Protocol: A Randomized Controlled Trial
Brief Title: Follicular Synchronization in PCOS Patients Undergoing ICSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Taman, lecturer, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R.19.07.557
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blinded clinical trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- • Study group (Active Comparator): It contains 100 patients will undergo ovarian stimulation with letrozole 2.5mg twice daily (Femara; Novartis Pharma Services, Basel, Switzerland) for 5 days starting from the first day of menstruation in combination with low dose step up stimulation with recombinant FSH starting in the third day of menstruation.
  Interventions: Drug: letrozole 2.5mg (Femara; Novartis Pharma Services, Basel, Switzerland)
- • Control group (No Intervention): It contains 100 patients will undergo ovarian stimulation with low dose step up stimulation with recombinant FSH starting in the third day of menstruation

INTERVENTIONS:
Drug: letrozole 2.5mg (Femara; Novartis Pharma Services, Basel, Switzerland) — letrozole /antagonist protocol
  Other Names: letroz 2.5mg (Sun Pharmaceuticals Industries Ltd.,India)
  Arms: • Study group

SUMMARY:
The use of GnRH antagonist protocol nowadays is the slandered protocol of controlled ovarian stimulation in patients with poly cystic ovarian syndrome (PCOS) because it decreases the incidence of OHSS(1, 2). However, this protocol may lead to asynchronous growth of follicles with an early dominant follicle specially in PCOS patients(3). In most of cases this phenomenon will affect the IVF outcomes(2, 4) Aromatase inhibitors (AIs) nowadays is recommended to be used for ovulation induction in patients with PCOS (5, 6).It has fewer side effects, and a shorter half-life than clomiphene citrate(CC), and no effect ON the endometrial receptivity. It is used in treating patients with chronic anovulation, unexplained infertility and poor ovarian reserve(7). It acts through decreasing estrogen levels and allows follicle stimulating hormone (FSH) release from the hypothalamus (8, 9). It could be used alone or with combination with human menopausal gonadotropin (HMG) specially in patients with CC resistant(10-13). It also improves the ovarian response to FSH when they are used in combination and it decreases the risk of OHSS (14).

This study aims to evaluate the effect of uses of letrozole in combination with HMG during ovarian stimulation in patients having PCOS undergoing IVF/ICSI on the follicular growth pattern, synchronized growth of follicles, maturity of oocyte and the quality of embryos.

DETAILED DESCRIPTION:
Participants in this study will be group of subfertile women undergoing IVF/ ICSI trial and having polycystic ovarian syndrome Inclusion criteria

1. Ages ≥20 and <40 years old
2. Women having the diagnosis of polycystic ovarian syndrome according to Rotterdam criteria (15)
3. Women who have at least one of the following indications for IVF or ICSI:

   1. Resistance to slandered ovulation induction and life style modification
   2. Tubal factors: unilateral or bilateral tubal obstruction, unilateral or bilateral salpingectomy or tubal ligation
   3. Male factors: oligoasthenozoospermia or obstructive azoospermia Exclusion criteria

1. Women with unexplained infertility. 2. women with poor ovarian reserve according to Bologna criteria (16). 3. Couples with known chromosomal abnormalities. 4. Women who refuse to participate in this study.

Methods

* patients will be randomly assigned into two groups (100 patients in each group): letrozole group (study group) and non letrozole group (control group). Treatment assignment will be blinded to patients, physicians, and nursing staff.
* All patients will receive combined oral pills before stimulation.
* letrozole 2.5mg twice daily (Femara; Novartis Pharma Services, Basel, Switzerland) will be given for 5 days starting from the second day of menstruation in combination with low dose step up stimulation with recombinant FSH in the study group.
* Allocated patients will be randomized into either of two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ages ≥20 and <40 years old 2. Women having the diagnosis of polycystic ovarian syndrome according to Rotterdam criteria (15) 3. Women who have at least one of the following indications for IVF or ICSI:

  1. Resistance to slandered ovulation induction and life style modification
  2. Tubal factors: unilateral or bilateral tubal obstruction, unilateral or bilateral salpingectomy or tubal ligation
  3. Male factors: oligoasthenozoospermia or obstructive azoospermia

Exclusion Criteria:

* 1. Women with unexplained infertility. 2. women with poor ovarian reserve according to Bologna criteria (16). 3. Couples with known chromosomal abnormalities. 4. Women who refuse to participate in this study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — subfertile women undergoing IVF/ ICSI trial and having polycystic ovarian syndrome
Enrollment: 200 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
the number of asynchronized follicles in both groups | 30 min
  • Asynchronization will considered when there is a difference of at least 2 mm between the dominant follicle and other follicles

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Taman, MD, Principal Investigator — Faculty of Medicine - Mansoura University
Locations (1):
- Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Inany HG, Youssef MA, Ayeleke RO, Brown J, Lam WS, Broekmans FJ. Gonadotrophin-releasing hormone antagonists for assisted reproductive technology. Cochrane Database Syst Rev. 2016 Apr 29;4(4):CD001750. doi: 10.1002/14651858.CD001750.pub4. PMID 27126581
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Hum Reprod. 2018 Sep 1;33(9):1602-1618. doi: 10.1093/humrep/dey256. PMID 30052961
- [Background] Wang R, Mol BW. The Rotterdam criteria for polycystic ovary syndrome: evidence-based criteria? Hum Reprod. 2017 Feb;32(2):261-264. doi: 10.1093/humrep/dew287. Epub 2016 Nov 9. PMID 28119448
- [Background] Ferraretti AP, Gianaroli L. The Bologna criteria for the definition of poor ovarian responders: is there a need for revision? Hum Reprod. 2014 Sep;29(9):1842-5. doi: 10.1093/humrep/deu139. Epub 2014 Jul 9. PMID 25008235
- [Background] Franik S, Eltrop SM, Kremer JA, Kiesel L, Farquhar C. Aromatase inhibitors (letrozole) for subfertile women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2018 May 24;5(5):CD010287. doi: 10.1002/14651858.CD010287.pub3. PMID 29797697
- [Background] Zhao Y, Ruan X, Mueck AO. Letrozole combined with low dose highly purified HMG for ovulation induction in clomiphene citrate-resistant infertile Chinese women with polycystic ovary syndrome: a prospective study. Gynecol Endocrinol. 2017 Jun;33(6):462-466. doi: 10.1080/09513590.2017.1292241. Epub 2017 Feb 28. PMID 28277124
- [Background] Wang R, Kim BV, van Wely M, Johnson NP, Costello MF, Zhang H, Ng EH, Legro RS, Bhattacharya S, Norman RJ, Mol BW. Treatment strategies for women with WHO group II anovulation: systematic review and network meta-analysis. BMJ. 2017 Jan 31;356:j138. doi: 10.1136/bmj.j138. PMID 28143834